CLINICAL TRIAL: NCT00225381
Title: Gas Kinetics and Metabolism in Anesthesia During Non Steady State
Status: Withdrawn | Type: Observational
Why Stopped: Non Applicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: R01 HL 42637 [HS# 2005-4256]; (UCI IRB ID)2005-4256 (Other: UC Irvine Institutional Review Board); R01HL042637 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Anesthetized Healthy Patients (ASA 1 or 2) in the Supine Position, Excluding Head, Neck and Head Surgeries; Anesthetized Patient With Severe Systemic Disease (ASA 3 or 4)
Keywords: Oxygen consumption; CO2 production; Indirect calorimetry; Non steady state; Anesthesia monitoring; Critical events during anesthesia; Acid base balance; Metabolism during anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- metabolic gas exchange and cardiac output
  Interventions: Device: connection of measuring device to anesthesia circuit; Procedure: placement of esophageal Doppler for cardiac output measurements; Device: Humidity sensor; Device: A mixing chamber (bymixer); Device: Pneumotachometer cuvette
- mass spectrometer and anaerobic metabolism
  Interventions: Device: connection of measuring device to anesthesia circuit; Procedure: drawing of blood sample through an arterial line, placed according to clinical criteria by primary anesthesia team; Device: Humidity sensor; Device: A mixing chamber (bymixer); Device: Pneumotachometer cuvette; Device: Mass spectrometer sampling port
- metaboic gas exchange and type of anesthesia induction
  Interventions: Device: connection of measuring device to anesthesia circuit; Device: Humidity sensor; Device: A mixing chamber (bymixer); Device: Pneumotachometer cuvette
- metabolic gas exchange and PEEP
  Interventions: Device: connection of measuring device to anesthesia circuit; Procedure: adding PEEP during anesthesia; Device: Humidity sensor; Device: A mixing chamber (bymixer); Device: Pneumotachometer cuvette
- metabolic gas exchange and trendelenburg position
  Interventions: Device: connection of measuring device to anesthesia circuit; Procedure: changing operating room bed position (head down and up position); Device: Humidity sensor; Device: A mixing chamber (bymixer); Device: Pneumotachometer cuvette
- Patients requiring tourniquet during surgery: Patients undergoing orthopaedic surgeries requiring tourniquet intervention. Oxygen consumption and CO2 production were measured before, during and after tourniquet release.
- Patients prone to metabolic acidosis: Oxygen consumption and CO2 measurements taken during long surgeries prone to metabolic acidosis.

INTERVENTIONS:
Device: connection of measuring device to anesthesia circuit — same as name
  Groups: mass spectrometer and anaerobic metabolism; metaboic gas exchange and type of anesthesia induction; metabolic gas exchange and PEEP; metabolic gas exchange and cardiac output; metabolic gas exchange and trendelenburg position
Procedure: drawing of blood sample through an arterial line, placed according to clinical criteria by primary anesthesia team — same
  Groups: mass spectrometer and anaerobic metabolism
Procedure: changing operating room bed position (head down and up position) — same
  Groups: metabolic gas exchange and trendelenburg position
Procedure: adding PEEP during anesthesia — same
  Groups: metabolic gas exchange and PEEP
Procedure: placement of esophageal Doppler for cardiac output measurements — same
  Groups: metabolic gas exchange and cardiac output
Device: Humidity sensor — Small conventional anesthesia T piece including tiny 2 thermometer inside
  Groups: mass spectrometer and anaerobic metabolism; metaboic gas exchange and type of anesthesia induction; metabolic gas exchange and PEEP; metabolic gas exchange and cardiac output; metabolic gas exchange and trendelenburg position
Device: A mixing chamber (bymixer) — 2 mixing chambers (bymixers) composed of 2 arms where one arm serves as a mixing (passive) arm for the measurement of mixed gas fraction. The bymixer is made of conventional anesthesia supplies and does not influence dead space nor circuit resistance.
  Groups: mass spectrometer and anaerobic metabolism; metaboic gas exchange and type of anesthesia induction; metabolic gas exchange and PEEP; metabolic gas exchange and cardiac output; metabolic gas exchange and trendelenburg position
Device: Pneumotachometer cuvette — The pneumotachometer cuvette is used by many anesthesia monitors to measure gas flow.
  Groups: mass spectrometer and anaerobic metabolism; metaboic gas exchange and type of anesthesia induction; metabolic gas exchange and PEEP; metabolic gas exchange and cardiac output; metabolic gas exchange and trendelenburg position
Device: Mass spectrometer sampling port — Designed for the anesthesia tubing and connected at the airway opening. it has small volume (3 mL) and do not influence circuit resistance.
  Other Names: V&F Instruments, Airsense (www.vandf.com)
  Groups: mass spectrometer and anaerobic metabolism

SUMMARY:
During clinical anesthesia, it is astonishing that CO2 monitoring consists mainly of end-tidal PCO2 to confirm endotracheal intubation and to estimate ventilation, and O2 monitoring consists of a single PO2 measurement to detect a hypoxic gas mixture. Better understanding of how O2 and CO2 kinetics monitoring can define systems pathophysiology will greatly enhance safety in anesthesia by detecting critical events such as abrupt decrease in cardiac output (Q.T) by vena-caval compression during abdominal surgery, occurrence of CO2 pulmonary embolism during laparoscopy, rising tissue O2 consumption (V.O2) during light anesthesia, and onset of anaerobic metabolism (V.CO2 is disproportionately higher than V.O2).

DETAILED DESCRIPTION:
During clinical anesthesia, it is astonishing that CO2 monitoring consists mainly of end-tidal PCO2 to confirm endotracheal intubation and to estimate ventilation, and O2 monitoring consists of a single PO2 measurement to detect a hypoxic gas mixture. Better understanding of how O2 and CO2 kinetics monitoring can define systems pathophysiology will greatly enhance safety in anesthesia by detecting critical events such as abrupt decrease in cardiac output (Q.T) by vena-caval compression during abdominal surgery, occurrence of CO2 pulmonary embolism during laparoscopy, rising tissue O2 consumption (V.O2) during light anesthesia, and onset of anaerobic metabolism (V.CO2 is disproportionately higher than V.O2).

In the previous grant period, discoveries of CO2 kinetics during non-steady state revealed significant gaps in understanding of O2 kinetics. To this end, a 5-compartment lung model of gas kinetics in the body during non-steady state has been developed, that incorporates complex interactions between O2 and CO2 in the lung, blood, and tissues. This computer model was used to formulate the following hypotheses, and will elucidate mechanisms underlying the subsequent measured data in anesthetized patients.

The investigators have already developed two innovative devices that are essential for the V.O2 measurement: A fast response temperature and humidity sensor, and a mixing device (a bymixer) for the measurement of mixed gas fraction, especially designed for anesthesia systems. The investigators have also designed a sophisticated bench system for the validation of both devices, which showed the high accuracy and performance of our measurements.

Hypotheses that will be tested in our overall research theme include:

* That pulmonary O2 uptake (V.O2) in anesthetized patients is much lower than the value quoted in the literature.
* That inhalation anesthesia influences V.O2 differently than total intravenous anesthesia (TIVA).
* That an acute decrease in cardiac output (Q.T) (by patient position change) will transiently decrease V.O2 but the decrease in CO2 elimination (V.CO2) is sustained because tissue CO2 stores are a hundred fold greater than O2 (please see previously approved IRB protocol, HS# 2000-1325).
* That positive end-expiratory pressure (PEEP) decreases V.O2 and V.CO2 due to decreases in Q.T and alveolar ventilation (V.A), and appearance of high ventilation-to-perfusion (V.A/Q.) units (please see previously approved IRB protocol, HS# 2000-1325).
* That Trendelenburg (head down) position increases V.O2 and V.CO2 due to increase in Q.T.
* That V.O2 can help to determine the necessity of blood transfusion.
* That the continuous measurement of the respiratory quotient (RQ=V.CO2/V.O2) can detect transition to anaerobic metabolism.
* That the continuous measurement of the respiratory RQ can be a good alternative to arterial blood gas sampling.
* That the continuous measurement of the respiratory RQ can determine the necessity of nutritional support during long operations.

In this protocol, the investigators will study the clinical implications of these measurements, believing that they are the missing links in anesthesia monitoring. Elucidating the mechanisms underlying this acute pathophysiology will advance the understanding of O2 and CO2 kinetics during non-steady state, and allow the non-invasive diagnosis of critical events during clinical anesthesia conferring increased safety, especially for the majority of healthy patients who receive only non-invasive monitoring.

A separate section of the study, which compliments the metabolic gas exchange study with the bymixer flow system is the examination of respiratory gas with a portable mass-spectrometer to detect volatile organic compounds during anaerobic metabolism. The experimental anaerobic model is adult patients undergoing a surgery that requires tourniquet. Anaerobic metabolism will be detected by acid base balance blood test, the bymixer flow measurement and the mass spectrometer. Anesthesia will be maintained by total intravenous anesthesia (TIVA) and each patient will have an arterial line. No other intervention would be taken. It is an observational type study.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients at UCIMC who are undergoing anesthesia and surgery are eligible for the studies
* Patients must be American Society of Anesthesiologists (ASA) Class 1 or 2 (generally healthy patients). We plan on studying 100 patients, divided into 5 equally numbered groups. A power analysis of the sample size shows the need for minimum of 20 patients. High risk 3 subgroups (ASA 3), approximately 20 adult patients (included within the 100 planned patients), will be investigated for the (1) RQ correlation with arterial blood gas, (2) for the exercise study and (3) for the esophageal Doppler studies. These study groups include patients that are categorized as ASA 1, 2 or 3, (total of 60 patients) however; the total number of ASA 3 patients will not exceed 20. Subjects having surgeries around the head and neck, as well as surgeries that require the patient to lie face down will be excluded from the study
* Gender and minority status will not be an exclusion factor for any potential study patient

Exclusion Criteria:

Cardiovascular:

* Significant vascular disease, especially cardiac and cerebral vascular disease
* Patients will be excluded if they have a history of having a myocardial infarction or cerebral vascular attack
* Significant hypertension (> 170 systolic, > 90 diastolic) (except for the high risk subgroup mentioned before)

Pulmonary:

* Significant asthma (mild persistent or greater according to the National Asthma Education and Prevention Program classification system) chronic obstructive pulmonary disease (COPD) (Stage II: Moderate COPD according to the Global Initiative for Chronic Obstructive Lung Disease classification
* Worsening airflow limitation, (FEV1 ≤30% ), and usually the progression of symptoms, with shortness of breath typically developing on exertion), bullous lung disease, or raised intra-cranial pressure (except for the high risk subgroup mentioned before)

Esophageal Doppler:

* If localized pathology is present, including pharyngeal tumor or significant esophageal varices, then the esophageal probe will not be used.

Emergency cases:

* Excluded from the study. Only elective patients will be enrolled.

Short surgeries:

* Surgeries that are expected to last 45 minutes or less will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients in the supine position excluding surgeries around the head and neck area
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2012-01-13 (Actual); Study Completion 2012-01-13 (Actual)

PRIMARY OUTCOMES:
Correlation between VO2 to type of anesthesia maintenance | 45 minutes
Correlation between acid base balance and indirect calorimetry | 2 hours
Detection of volatile organic compound during anaerobic metabolism | 3 hours
Influence of anesthesia induction on metabolic gas exchange | 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Breen, MD, FRCPC, Principal Investigator — UCI Medical Center; Abraham Rosenbaum, MD, Study Director — UCI Medical Center
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Rosenbaum A, Kirby C, Breen PH. Measurement of oxygen uptake and carbon dioxide elimination using the bymixer: validation in a metabolic lung simulator. Anesthesiology. 2004 Jun;100(6):1427-37. doi: 10.1097/00000542-200406000-00015. PMID 15166562
- [Background] Rosenbaum A, Breen PH. Novel, adjustable, clinical bymixer measures mixed expired gas concentrations in anesthesia circle circuit. Anesth Analg. 2003 Nov;97(5):1414-1420. doi: 10.1213/01.ANE.0000083420.15268.3A. PMID 14570659
- [Background] Breen PH, Isserles SA, Taitelman UZ. Non-steady state monitoring by respiratory gas exchange. J Clin Monit Comput. 2000;16(5-6):351-60. doi: 10.1023/a:1011447500984. PMID 12580218
- [Background] Breen PH. Importance of temperature and humidity in the measurement of pulmonary oxygen uptake per breath during anesthesia. Ann Biomed Eng. 2000 Sep;28(9):1159-64. doi: 10.1114/1.1312184. PMID 11132200
- [Background] Breen PH, Serina ER. Bymixer provides on-line calibration of measurement of CO2 volume exhaled per breath. Ann Biomed Eng. 1997 Jan-Feb;25(1):164-71. doi: 10.1007/BF02738547. PMID 9124730
- [Background] Breen PH, Serina ER, Barker SJ. Measurement of pulmonary CO2 elimination must exclude inspired CO2 measured at the capnometer sampling site. J Clin Monit. 1996 May;12(3):231-6. doi: 10.1007/BF00857644. PMID 8823647
- [Background] Breen PH, Mazumdar B, Skinner SC. Capnometer transport delay: measurement and clinical implications. Anesth Analg. 1994 Mar;78(3):584-6. doi: 10.1213/00000539-199403000-00027. PMID 8109779
- [Background] Breen PH, Isserles SA, Harrison BA, Roizen MF. Simple computer measurement of pulmonary VCO2 per breath. J Appl Physiol (1985). 1992 May;72(5):2029-35. doi: 10.1152/jappl.1992.72.5.2029. PMID 1601815
- [Background] Isserles SA, Breen PH. Can changes in end-tidal PCO2 measure changes in cardiac output? Anesth Analg. 1991 Dec;73(6):808-14. doi: 10.1213/00000539-199112000-00023. PMID 1952183
- [Result] Rosenbaum A, Breen PH. Importance and interpretation of fast-response airway hygrometry during ventilation of anesthetized patients. J Clin Monit Comput. 2007 Jun;21(3):137-46. doi: 10.1007/s10877-006-9065-5. Epub 2007 Mar 16. PMID 17364215
- [Result] Rosenbaum A, Kirby C, Breen PH. New metabolic lung simulator: development, description, and validation. J Clin Monit Comput. 2007 Apr;21(2):71-82. doi: 10.1007/s10877-006-9058-4. Epub 2007 Mar 1. PMID 17333487
- See also: Related Info — http://www.anesthesiology.uci.edu/research.shtml